CLINICAL TRIAL: NCT01451216
Title: The Evaluation of Balance Control by Quantification of the Temporospatial Measures of Functional Reach Test
Brief Title: The Evaluation of Balance Control by Quantification of Temporospatial Measures While Forward and Side Reaching
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ofer Keren, Dr. Ofer Keren, Sheba Medical Center
Other Study IDs: SHEBA-11-8745-OK-CTIL
Record Dates: First submitted 2011-10-10; First posted 2011-10-13 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Brain Injury
Keywords: Acquired brain injury; Balance control; Functional reach
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ABI 50-70 y: patients suffering from acquired brain injury aged 50-70 years old
- ABI 25-50y: Patients suffering from acquired brain injury aged 25-50 years oled

SUMMARY:
Balance control is the sum action of the sense and reaction systems. In order to perform different activities in different postures one must have the ability to control and to adjust his balance in different conditions.A deficit in brain action following injury, disease or aging can undermine the ability to control balance and increase the risk to fall.The limitation in gait and mobility can increase morbidity. There is a limited number of tools evaluating and recording balance control ability. Most of this tools are observational and can be used in the clinical field. The aim of this work is to estimate the feasibility of an objective tool that can evaluate balance by tracking objective quantitative measures during the standard physical therapy session without using an expensive equipment. By using this tool the therapist can monitor the patient and collect quantitive data while performing tasks while keeping balance. This tool will allow the therapist to detect changes in balance and evaluate the effect of different conditions on the patients balance. This tool is based on the well known functional reach test. The addition of this tool to the test is the use of a simple camera and a computer softwear that will collect the data and analyze it while performing the test. This tool will give the therapist information on the responsiveness and the spatiotemporal measures of the performance. The aim of this work is to check what is the contribution of spatiotemporal measures of the functional reach test among patients suffering from acquired brain injury to the understanding of the motor function and balance control of people suffering from brain injury. .

ELIGIBILITY:
Inclusion Criteria:

* Acquired Brain Injury patients Can stand without assistance for at list 10 sec. Can walk 10m with or without walking aid Has no limitation in RPOM of the upper or lower limb need no guardian

Exclusion Criteria:

* Apraxia of all kind Aphasia Neglect

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acquired Brain patients who are hospitalized in the Brain Injury department in Sheba Medical Center Israel for rehabilitation. Males and females, from them 20 aged 25-50, 20 aged 50-70.All the participents are able to stand without assistance for at list 10 sec. and can walk with or without walking aid. In addition they will not have any limitation of the upper or lower limbs range of motion.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-11

CONTACTS AND LOCATIONS:
Overall Officials: Michal Katz-Leurar, PhD, Study Chair — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel